CLINICAL TRIAL: NCT05439174
Title: Impact of Intradialytic Parenteral Nutrition on Nutrition Markers in Patients Receiving In-Center Hemodialysis
Brief Title: Impact of IDPN on Nutrition Markers in Patients Receiving ICHD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Patient Care America (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IDPN and ICHD Study Protocol
Record Dates: First submitted 2022-06-23; First posted 2022-06-30 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: End-stage Renal Disease; Malnutrition; Protein
MeSH Terms: conditions — Kidney Failure, Chronic; Kwashiorkor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intradialytic Parenteral Nutrition — Intradialytic parenteral nutrition (IDPN) is compounded using a combination of dextrose (D70%) and amino acids (Prosol 20%, Clinisol 15%, or Plenamine 15%) with the option of adding lipids (Intralipid 20% prior to 8/2020, Clinolipid starting 8/2020 and after).
  Each prescription is dosed based on patient height, weight, and other nutrition considerations including but not limited to presence of wounds, recent hospitalizations, electrolyte imbalance, etc. Adjustments to prescription are made on an as needed basis to increase or decrease goal infusion rate, adjust protein levels, and/or add or remove lipids.
  Other Names: NutriRite

SUMMARY:
Evaluate the impact of intradialytic parenteral nutrition (IDPN) compounded with Clinisol, Prosol, and/or Clinolipid on albumin levels and weight in patients with end-stage renal disease (ESRD) undergoing in-center hemodialysis. Determine the average duration of time it takes for albumin levels to rise ≥0.2g/dL from the initiation of IDPN therapy as this has been associated with significant change in mortality and hospitalization risk. The investigators expect levels to rise significantly within 4-6 months, there may be a difference in outcome in patients receiving IDPN compounded with amino acids and dextrose only vs IDPN compounded with amino acids, lipid, and dextrose.

DETAILED DESCRIPTION:
Intradialytic parenteral nutrition (IDPN) has been identified as a means of improving nutrition status in malnourished hemodialysis patients who cannot meet calorie and protein needs with oral intake alone. The retrospective chart review spanning 3 years will be conducted on in-center hemodialysis patients receiving IDPN concurrent with their dialysis treatment. This study will evaluate the impact of intradialytic parenteral nutrition (IDPN) compounded with Clinisol, Prosol, Plenamine, Intralipid and/or Clinolipid on albumin levels in patients with end-stage renal disease (ESRD) undergoing in-center hemodialysis and determine if addition of Clinolipid changes response to IDPN therapy compared to IDPN without lipids or IDPN with Intralipid. The primary endpoint is change in albumin levels from baseline (average albumin of up to 3 months prior to initiation of IDPN therapy) to 6 months after IDPN therapy initiation for the full analysis set. Secondary endpoints will be analyzed and include: distinguishing factors between those that respond to IDPN therapy (0.2g/dL or more increase in albumin levels) and those that do not; assessing time to IDPN response (increase of 0.2g/dL in albumin levels); determining factors that predict IDPN response; and comparing amount of change in albumin levels, percent of patients responding to IDPN therapy, and amount of time to IDPN response between those that receive lipids with IDPN therapy and those that do not receive lipids.

ELIGIBILITY:
Inclusion Criteria:

* Receiving in-center hemodialysis 3 days per week
* Having any diagnosis of ESRD
* ICD-10 code N18.6
* IDPN therapy initiated between May 1, 2018 and April 30, 2021 (evaluating through October 31, 2021)
* Baseline data available, average of up to 3 months of albumin levels available prior to start of therapy
* Age 18 years or older at IDPN therapy initiation
* Consented to have their medical records used for research

Exclusion Criteria:

* - Dialysis prescription deviates from the standard 3 days per week
* IDPN or intraperitoneal nutrition (IPN) therapy was initiated outside the research window
* Under 18 years of age at IDPN initiation
* History of liver disease or gastric bypass
* Undergoing cancer treatment at any time during IDPN therapy
* Receiving enteral nutrition support or total parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all adult (18 years or older) patients with end-stage renal disease (ESRD) receiving IDPN therapy while undergoing in-center hemodialysis 3 days per week.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Time from baseline to clinically significant improvement in albumin | 6 months
  Albumin levels of study population will rise significantly (0.2g/dL) after 6 months of intradialytic parenteral nutrition (IDPN) therapy

SECONDARY OUTCOMES:
Difference between use of IDPN without lipids, with Clinolipid, and with Intralipid | 6 months
  Response time to therapy over an observation period of 6 months will be improved in patients receiving IDPN compounded with Clinolipid compared to patients receiving IDPN with Intralipid or no lipids.

CONTACTS AND LOCATIONS:
Locations (1):
- Patient Care America, Pompano Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shah A, Bross R, Shapiro BB, Morrison G, Kopple JD. Dietary energy requirements in relatively healthy maintenance hemodialysis patients estimated from long-term metabolic studies. Am J Clin Nutr. 2016 Mar;103(3):757-65. doi: 10.3945/ajcn.115.112995. Epub 2016 Feb 10. PMID 26864370
- [Background] Carrero JJ, Thomas F, Nagy K, Arogundade F, Avesani CM, Chan M, Chmielewski M, Cordeiro AC, Espinosa-Cuevas A, Fiaccadori E, Guebre-Egziabher F, Hand RK, Hung AM, Ikizler TA, Johansson LR, Kalantar-Zadeh K, Karupaiah T, Lindholm B, Marckmann P, Mafra D, Parekh RS, Park J, Russo S, Saxena A, Sezer S, Teta D, Ter Wee PM, Verseput C, Wang AYM, Xu H, Lu Y, Molnar MZ, Kovesdy CP. Global Prevalence of Protein-Energy Wasting in Kidney Disease: A Meta-analysis of Contemporary Observational Studies From the International Society of Renal Nutrition and Metabolism. J Ren Nutr. 2018 Nov;28(6):380-392. doi: 10.1053/j.jrn.2018.08.006. PMID 30348259
- [Result] Marsen TA, Beer J, Mann H; German IDPN-Trial group. Intradialytic parenteral nutrition in maintenance hemodialysis patients suffering from protein-energy wasting. Results of a multicenter, open, prospective, randomized trial. Clin Nutr. 2017 Feb;36(1):107-117. doi: 10.1016/j.clnu.2015.11.016. Epub 2015 Dec 12. PMID 26708726
- [Result] Pupim LB, Flakoll PJ, Ikizler TA. Nutritional supplementation acutely increases albumin fractional synthetic rate in chronic hemodialysis patients. J Am Soc Nephrol. 2004 Jul;15(7):1920-6. doi: 10.1097/01.asn.0000128969.86268.c0. PMID 15213282
- [Result] Pupim LB, Flakoll PJ, Brouillette JR, Levenhagen DK, Hakim RM, Ikizler TA. Intradialytic parenteral nutrition improves protein and energy homeostasis in chronic hemodialysis patients. J Clin Invest. 2002 Aug;110(4):483-92. doi: 10.1172/JCI15449. PMID 12189242
- [Result] Ortiz-Ortiz L, Contreras MF, Bojalil LF. The assay of delayed hypersensitivity to ribosomal proteins from Nocardia. Sabouraudia. 1972 Jul;10(2):147-51. doi: 10.1080/00362177285190291. No abstract available. PMID 4557877